CLINICAL TRIAL: NCT02531685
Title: A Phase 1 Double-Blind Placebo-Control Dose Escalating Study to Evaluate the Safety and Immunogenicity of Double Mutant Heat-Labile Toxin LTR192G/L211A (dmLT) From Enterotoxigenic Escherichia Coli (ETEC) by Intradermal (ID) Vaccination in Healthy Adults
Brief Title: Phase 1 Study of dmLT ID Vaccination in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 13-0013; HHSN272201300022I
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10-20

CONDITIONS: Gastroenteritis Escherichia Coli
Keywords: dmLT; Enteric; Escherichia coli Infections; Shigella; Toxin LTR192G/L211A
MeSH Terms: conditions — Escherichia coli Infections; Dysentery, Bacillary | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): 13 subjects receive 0.1 mcg dmLT intradermally on days 1, 22 and 43. 3 subjects receive placebo.
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 2 (Experimental): 13 subjects receive 0.3 mcg dmLT intradermally on days 1, 22 and 43. 3 subjects receive placebo.
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 3 (Experimental): 13 subjects receive 1.0 mcg dmLT intradermally on days 1, 22 and 43. 3 subjects receive placebo.
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 4 (Experimental): A sentinel group of 5 subjects receive 2.0 mcg dmLT intradermally on days 1, 22, and 43. 1 subject receives placebo.
  Safety data from days 1-14 in sentinel will be reviewed and upon approval to proceed, 8 additional subjects receive 2.0 mcg dmLT intradermally on days 1, 22 and 43. 2 subjects receive placebo.
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 5 (Experimental): Up to 31 subjects receive TBD mcg dmLT intradermally on days 1, 22 and 43. 4 subjects receive placebo.
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine

INTERVENTIONS:
Other: Placebo — Placebo: 0.9% Sodium Chloride injection.
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — LT(R192G/L211A), or dmLT is formulated as a freeze-dried (lyophilized), white to off-white cake, containing 700mcg of vaccine protein in a 3 ml, multi-dose.

SUMMARY:
This study is to determine the safety and immunogenicity of an Enterotoxigenic Escherichia coli (ETEC) candidate vaccine, attenuated recombinant Double Mutant Heat-Labile Toxin (dmLT) from ETEC, administered by the Intradermal (ID) route. The sample size has been determined based on the historic sample, not on power calculations.The study will involve 99 subjects (83 vaccinees and 16 placebo controls) in 4 consecutive cohorts of 16 individuals each (13 vaccinees and 3 placebo controls) and the final cohort of 35 (31 vaccinees and 4 placebos) subjects. The primary objective is to assess the safety and tolerability of dmLT vaccine when administered in three doses intradermally over a range of dosages in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, single site outpatient Phase 1 study in healthy adults to determine the safety and immunogenicity of an Enterotoxigenic Escherichia coli (ETEC) candidate vaccine, attenuated recombinant Double Mutant Heat-Labile Toxin (dmLT) from ETEC, administered by the Intradermal (ID) route. The sample size has been determined based on the historic sample, not on power calculations.The study will involve 99 subjects (83 vaccinees and 16 placebo controls) in 4 consecutive cohorts of 16 individuals each (13 vaccinees and 3 placebo controls) and the final cohort of 35 (31 vaccinees and 4 placebos) subjects. A total of 16 subjects (to retain 10 vaccinees and 1 placebo evaluable subjects) in each cohort 1-4 will initially be recruited, 13 subjects each will receive three separate doses of dmLT intradermally at 1, 22 and 43-day, and 3 subjects in each cohort will receive three doses of a placebo (saline) in a blinded fashion. Because of concerns of local reactogencity in cohort 3, cohort 4 will include a sentinel group of 6 subjects that is assessed prior to dosing the remaining 10 subjects. Proceeding to the remaining subjects will be based on review of safety data obtained from days 1-14 after the first dose in the sentinel subjects by the ISM, PI and MM. As this is an outpatient study, subjects will receive their vaccinations and remain in clinic for observation for a minimum of 30 minutes. Safety data will be reviewed by Safety Monitoring Team or Committee. Subjects may be replaced to ensure 10 evaluable subjects in each single cohort, as defined by receiving all 3 vaccine doses. If replacement subjects will be included if needed and they will be randomized per cohort as a single group to include 1 subject to receive placebo to maintain the blind and ensure there are one placebos in each cohort. Final confirmatory cohort will include up to 35 vaccinees randomly selected to receive either 1, 2 or 3 vaccine doses or placebo. The study duration is approximately 1.5-2 years, including 6 months of follow-up and approximately 9 months for subject duration. The primary objective is to assess the safety and tolerability of dmLT vaccine when administered in three intradermal doses over a range of dosages levels in healthy adult subjects. The secondary objectives are: 1. To assess long-term safety follow-up from immunization through 6 months post last vaccination; 2. Following ID administration of dmLT vaccine over a range of dosages levels evaluate dmLT-specific immune response by assays.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18-45, inclusive.
2. Provide written informed consent before initiation of any study procedures.
3. Are in general good health.

   * As defined by being without:
   * significant medical illness,

     * clinically significant physical examination findings, including vitals, as determined by the PI, and ---screening laboratory values outside the site's normal limits.
4. Within 46 days of vaccination, have normal screening laboratories.

   -Screening labs include white blood cells (WBCs) , hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), sodium, potassium, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST).
5. Have normal screening laboratories for urine protein. Trace protein is acceptable.
6. Hemoglobin (Hgb) A1C < 6.5 percent at screening.
7. Agrees to complete all study visits and procedures and to provide a screening stool sample.
8. Female subjects must be of non-childbearing potential or if of childbearing potential, must be using an effective method of birth control or must be abstinent.

   -Non-childbearing potential is defined as surgically sterile or postmenopausal for > one year.

   --Effective methods of birth control include the use of hormonal or barrier birth control such as implants, injectable contraceptives, combined oral contraceptives, intrauterine devices [IUDs], cervical sponges, diaphragms, or condoms with spermicidal agents within 2 months of vaccination. Female subjects must be using an effective method of birth control or practice abstinence and must agree to continue such precautions during the study and for 30 days after the Day 43 study visit.

   ---A woman is eligible if she is monogamous with a vasectomized male.
9. Male subjects must agree not to father a child for 30 days after the last dose of the vaccine.
10. Agrees not to participate in another clinical trial during the study period.
11. Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine.
12. Potential subjects must be willing to adhere to the following prohibitions and restrictions on exercise during the course of the study to be eligible for participation.

    * Strenuous exercise (e.g., long distance running > 5km/day, weight lifting, or any physical activity to which the subject is not accustomed) is to be avoided for at least 72 hours prior to each study drug administration (and the Follow-up visit).

Exclusion Criteria:

1. Women who are pregnant or lactating or have a positive serum pregnancy test at screening or positive urine pregnancy test on vaccination days.
2. Abnormal vital signs, defined as:

   -Hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days.

   --Palpated heart rate < 55 or > 100 beats/minute at rest on 2 separate days.

   ---If heart rate between 45 and 55, subjects may be enrolled with an EKG that demonstrates normal sinus rhythm and does not document conduction disorders.

   ----Oral Temperature >= 38.0 Degrees Celsius (100.4 Degrees Fahrenheit).
3. Symptoms of an acute self-limited illness, including an oral temperature >= 38.0 Degrees Celsius (100.4 Degrees Fahrenheit), such as an upper respiratory infection or gastroenteritis within 7 days of administration of Double Mutant Heat-Labile Toxin (dmLT).
4. Positive hepatitis C, or Human Immunodeficiency Virus (HIV) serology or positive hepatitis B serology not consistent with prior hepatitis B immunization.
5. Have a positive urine drug screen for opiates.
6. History of antimicrobial treatment in the 2 weeks before any administration of dmLT.
7. Received previous experimental E. coli, Labile Toxin (LT), or cholera vaccines or live E. coli or Vibrio cholera challenges; or previous known infections with cholera or diarrheagenic E. coli.
8. Abnormal routine bowel habits as defined by fewer than three stools per week or more than two stools per day in the past 6 months.
9. History of chronic gastrointestinal illness.

   -This includes severe dyspepsia (mild or moderate heartburn or epigastric pain occurring no more than three times per week is permitted), or other significant gastrointestinal tract disease.
10. Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy.
11. History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy.
12. Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (> 800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months.
13. Long-term use is defined as longer than 14 days. Nasal and topical steroids are allowed.

    -Long-term use is defined as longer than 14 days. Nasal and topical steroids are allowed.
14. Have a diagnosis of schizophrenia or other major psychiatric diagnosis.
15. Are receiving impermissible psychiatric drugs.

    -The following psychiatric drugs are not permitted: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, or lithium citrate.

    --Subjects who are receiving a single antidepressant drug and are stable for at least 3 months before enrollment without de-compensating symptoms are allowed to be enrolled in the study.
16. History of receiving Immunoglobulin (Ig) or other blood product within the 3 months before enrollment in this study.
17. Subjects who have traveled to an ETEC-endemic area within the past 3 years or have been raised in a cholera or ETEC endemic area.

    -Defined as Africa, Middle East, South Asia, or Central or South America.
18. Subjects who plan to travel to an ETEC-endemic area during the long-term safety follow-up period (6 months after last vaccination) of the study.

    -Defined as Africa, Middle East, South Asia, or Central or South America.
19. Received any licensed vaccine prior to enrollment in this study or plans to receive any licensed vaccine after any study vaccination.

    -Inactivated vaccines may not have been received within 2 weeks of enrollment or within 2 weeks after any study vaccination. Live vaccines may not have been received within 4 weeks of enrollment, while on study, or within 4 weeks of final study visit.
20. An acute or chronic medical condition that, in the opinion of the investigator, would render administration of dmLT unsafe or would interfere with the evaluation of responses. -This includes, but is not limited to: known or suspected immunodeficiency, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, history of diabetes, cancer (other than a healed skin lesion), heart disease (in the hospital for a heart attack, history of irregular heart beat or have had postural hypotension in the past year, unconsciousness (other than a single brief concussion), seizures (other than with fever when subject was a child <5 years old), asthma requiring treatment with inhaler or medication in the prior 2 years, autoimmune disease or eating disorder, and transplant recipients.
21. Have received experimental products within 30 days prior to study entry or plan to receive experimental products at any time during the study.
22. History of alcohol or drug abuse in the last 5 years.
23. Plans to travel outside of the USA in the time between study vaccination and 4 weeks following the final vaccination.
24. Any condition that would, in the opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
25. Use of prescription or over-the-counter (OTC) anti-inflammatory medications 48 hours prior to receiving the investigational product.

    -This includes medications that contain naproxen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs.
26. Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.
27. Known allergies to study compound or components of the study vaccine.
28. Special populations, e.g., non-English speakers, children, illiterate or non-writing individuals, vulnerable populations.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events (AEs) | 7 Days following each vaccination
Occurrence of vaccine-related, non-solicited adverse events (AEs) | Day 1 through 30 days following last vaccination

SECONDARY OUTCOMES:
Occurrence of vaccine-related serious adverse events (SAEs) | Day 1 through 6 months following last vaccination
Occurrence of vaccine-related, non-solicited adverse events (AEs) | Day 1 through 6 months after last vaccination
Proportion of subjects with > / = 2-fold rise from the baseline in double mutant heat-labile toxin (dmLT)-specific toxin neutralization IgA-ALS titers at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > / = 2-fold rise from the baseline in double mutant heat-labile toxin (dmLT)-specific toxin neutralization IgG-ALS titers at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > / = 4 fold rise from the baseline double mutant heat-labile toxin (dmLT)-specific fecal IgA titers at any time | Day 1 through 8 days (cohorts 5A and 5B) or 29 days (cohorts 1-4 and 5C) following last vaccination
Proportion of subjects with > / = 4 fold rise from the baseline ratio of antigen-specific IgA over total IgA at any time | Day 1 through 8 days (cohorts 5A and 5B) or 29 days (cohorts 1-4 and 5C) following last vaccination
Proportion of subjects with > / = 4-fold rise from the baseline in double mutant heat-labile toxin (dmLT)-specific serum IgA titers at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > / = 4-fold rise from the baseline in double mutant heat-labile toxin (dmLT)-specific serum IgG titers at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > / = 4-fold rise from the baseline in the ratio of double mutant heat-labile toxin (dmLT)-specific toxin neutralization titer at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > 8 IgA-ASC/10^6 peripheral blood mononuclear cells (PBMCs) at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with > 8 IgG-ASC/10^6 peripheral blood mononuclear cells (PBMCs) at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
Proportion of subjects with B or T cell memory at any time | Day 1 through 56 days (Cohorts 1-4) or 6 months (Cohort 5) following last vaccination
  Determined by EliSpot
Proportion of subjects with IgA double mutant heat-labile toxin (dmLT)-specific circulating ASC expressing gut homing receptors (integrin alpha4beta7 in the absence or presence of CD62L) at any time in cohort 5 only | 8 days following first vaccination through 8 days following last vaccination
Proportion of subjects with IgG double mutant heat-labile toxin (dmLT)-specific circulating ASC expressing gut homing receptors (integrin alpha4beta7 in the absence or presence of CD62L) at any time in cohort 5 only | 8 days following first vaccination through 8 days following last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Pasetti MF, Milletich PL, White JA, Butts J, Brady RC, Dickey MD, Ballou C, Maier N, Sztein MB, Baqar S, Louis Bourgeois A, Bernstein DI. Safety and immunogenicity in humans of enterotoxigenic Escherichia coli double mutant heat-labile toxin administered intradermally. NPJ Vaccines. 2025 Feb 1;10(1):23. doi: 10.1038/s41541-025-01071-7. PMID 39893179